CLINICAL TRIAL: NCT07120308
Title: An Investigator-initiated Single-center, Randomized, Double-blind, Placebo-controlled Clinical Study Evaluating the Efficacy and Safety of ZKY001 Eye Drops in the Treatment of Corneal Epithelial Defects Caused by Neurotrophic Keratitis
Brief Title: To Evaluate the Efficacy and Safety of ZKY001 Eye Drops in the Treatment of Corneal Epithelial Defects Caused by Neurotrophic Keratitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhaoke (Guangzhou) Ophthalmology Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIT2021-ZKY001-NK
Record Dates: First submitted 2021-09-16; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Corneal Epithelial Defect

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0.002% ZKY001 eye drops（Herpes simplex keratitis group） (Experimental): NK caused by Herpes simplex keratitis 0.002% ZKY001 eye drops，1 drop each time, 4 times a day. Start on D1, continuously for 56±3 days. It is recommended that the eye drops be taken at intervals of 4 to 6 hours.
  Interventions: Drug: ZKY001 eye drops
- Vehicle（Herpes simplex keratitis group） (Placebo Comparator): NK caused by Herpes simplex keratitis Vehicle，1 drop each time, 4 times a day. Start on D1, continuously for 56±3 days. It is recommended that the eye drops be taken at intervals of 4 to 6 hours.
  Interventions: Drug: Vehicle (placebo)
- 0.002% ZKY001 eye drops（Diabetes group） (Experimental): NK caused by diabetes 0.002% ZKY001 eye drops,1 drop each time, 4 times a day. Start on D1, continuously for 56±3 days. It is recommended that the eye drops be taken at intervals of 4 to 6 hours.
  Interventions: Drug: ZKY001 eye drops
- Vehicle（Diabetes group） (Placebo Comparator): NK caused by diabetes Vehicle，1 drop each time, 4 times a day. Start on D1, continuously for 56±3 days. It is recommended that the eye drops be taken at intervals of 4 to 6 hours.
  Interventions: Drug: Vehicle (placebo)

INTERVENTIONS:
Drug: ZKY001 eye drops — Administer to eyes
  Arms: 0.002% ZKY001 eye drops（Diabetes group）; 0.002% ZKY001 eye drops（Herpes simplex keratitis group）
Drug: Vehicle (placebo) — Administer to eyes
  Arms: Vehicle（Diabetes group）; Vehicle（Herpes simplex keratitis group）

SUMMARY:
An investigator-initiated single-center, randomized, double-blind, placebo-controlled clinical study .The main purpose is to evaluate the effectiveness of ZKY001 eye drops in treating corneal epithelial defects caused by neurotrophic keratitis in patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 years ≤ aged ≤ 80 years； Consistent with the diagnosis of neurotrophic keratitis caused by diabetes or the herpes simplex virus； Patients with Stage 2 or Stage 3 neurotrophic keratitis，involving only one eye； PED or corneal ulceration of at least 2 weeks' duration refractory to one or more conventional non-surgical treatments for neurotrophic keratitis (e.g., preservative-free artificial tears, gels or ointments; discontinuation of preserved topical drops； medications that can decrease corneal sensitivity; therapeutic contact lenses and Cenegermin eye drops)； Signed informed consent forms。

Exclusion Criteria:

* Patients with Stage 2 or 3 NK affecting both eyes； Any active ocular infection (bacterial, viral, fungal or protozoal) or active ocular inflammation not related to NK in the affected eye； Any other ocular disease requiring topical ocular treatment in the affected eye during the study treatment period； Patients with severe vision loss in the affected eye with no potential for visual improvement in the opinion of the Investigator because of the study treatment； Schirmer's test without anesthesia ≤ 3 mm/ 5 minutes in the affected eye； Patients with severe blepharitis and/or severe meibomian gland disease in the affected eye； History of laser surgical procedures in the affected eye within the 3 months before study enrollment，history of any ocular surgery (except retinal laser photocoagulation) in the affected eye within the 1 month before study enrollment. No ocular surgery (except retinal laser photocoagulation) will be performed on the affected eye during the study period； Prior surgical procedure(s) for the treatment of NK (e.g., complete tarsorrhaphy, conjunctival flap, etc.) in the affected eye except for amniotic membrane transplantation could only be enrolled 2 weeks after the membrane had disappeared within the area of the PED or corneal ulcer or at least 6 weeks after the date of the amniotic membrane transplantation procedure； Use of therapeutic contact lenses or contact lens wear for refractive correction during the study treatment periods in the eye with NK； Anticipated need for obliteration lacrimal punctum during the study treatment period. Patients with obliteration lacrimal punctum or lacrimal plugs inserted prior to the study were eligible for enrollment if the obliteration lacrimal punctum was maintained during the study； Evidence of corneal ulceration involving the posterior third of the corneal stroma, corneal melting or perforation in the affected eye； Presence or history of any ocular or systemic disorder or condition that may hinder the efficacy of the study treatment or its evaluation, could possibly have interfered with the interpretation of study results, or could have been judged by the Investigator to be incompatible with the study visit schedule or conduct (e.g., progressive or degenerative corneal or retinal conditions, uveitis, optic neuritis, poorly controlled diabetes, autoimmune disease, systemic infection, neoplastic diseases)； Any need for or anticipated change in the dose of systemic medications known to impair the function of the trigeminal nerve (e.g., neuroleptics, antipsychotic and antihistamine drugs). These treatments were allowed during the study if initiated prior to 30 days before study enrollment on condition that treatment remains stable throughout the course of the study treatment period； Known hypersensitivity to one of the components of the study or procedural medications (e.g., fluorescein)； History of drug, medication or alcohol abuse or addiction； Participation in another clinical study at the same time as the present study；

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with corneal epithelial healing（<0.5 mm lesion size） at D57. | Day 57
  corneal epithelial healing（<0.5 mm lesion size）

SECONDARY OUTCOMES:
Duration of corneal healing (<0.5 mm lesion size). | D57
  corneal healing (<0.5 mm lesion size).
Percentage of improvement in corneal epithelial defect from baseline at D29、D57 | D29、D57
  improvement in corneal epithelial defect
Improvement in corneal fluorescein staining scores from baseline at D29、D57 | D29、D57
  Improvement in corneal fluorescein staining scores
Improvement in corneal sensitivity from baseline at D29、D57 | D29、D57
  Improvement in corneal sensitivity

CONTACTS AND LOCATIONS:
Locations (1):
- Xiamen Eye Center of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No